CLINICAL TRIAL: NCT05778786
Title: Design Validation of Toric Contact Lenses in Senofilcon A With a Blue-Blocking Chromophore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6521
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to wear bilaterally two different study lenses, one at a time, for a minimum of 8 hours per day for at least 5 days during each wear period, over two wear periods (test then control) with a washout period of 7+/-2 days duration between wear periods.
  Interventions: Device: Acuvue Oasys 1 Day for Astigmatism; Device: TRA100/TRA200 series toric contact lens with HEVL-blocking chromophore
- Control/Test (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Control/Test sequence, to wear bilaterally two different study lenses, one at a time, for a minimum of 8 hours per day for at least 5 days during each wear period, over two wear periods (control then test) with a washout period of 7+/-2 days duration between wear periods.
  Interventions: Device: Acuvue Oasys 1 Day for Astigmatism; Device: TRA100/TRA200 series toric contact lens with HEVL-blocking chromophore

INTERVENTIONS:
Device: Acuvue Oasys 1 Day for Astigmatism — CONTROL
Device: TRA100/TRA200 series toric contact lens with HEVL-blocking chromophore — TEST

SUMMARY:
This will be a 4-visit, randomized, controlled, single-masked, bilateral wear, dispensing, 2-treatment, 2-sequence, 2-period crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 years of age (inclusive) at the time of screening.
4. Habitually wear soft contact lenses in both eyes in a daily or daily disposable wear modality (i.e., not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past four weeks.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study:

   1. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps
   2. Cylinder powers (DC) -0.75 and -1.25
   3. Axes (°) 170, 180, 10, 80, 90, 100
7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have an ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (10):
- United States (10):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Omega Vision Center, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Optometry Group, LLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 188 subjects were enrolled in this study. All 188 enrolled subjects were dispensed at least one study lens. Of those dispensed, 179 subjects completed the study while 9 subjects were discontinued.
Groups:
- Test-senofilcon A (C3)/Control-senofilcon A (C3): Subjects in this arm were randomized to receive the Test lens during the first period of the study and the Control lens during the second period of the study.
- Control-senofilcon A (C3)/ Test-senofilcon A (C3): Subjects in this arm were randomized to receive the Control lens during the first period of the study and the Test lens during the second period of the study.
Period: Period 1
Arm/Group | Test-senofilcon A (C3)/Control-senofilcon A (C3) | Control-senofilcon A (C3)/ Test-senofilcon A (C3)
Started | 95 | 93
Completed | 91 | 90
Not Completed | 4 | 3
Not completed — COVID-19 Related | 3 | 3
Not completed — Withdrew Consent during Study | 1 | 0
Period: Period 2
Arm/Group | Test-senofilcon A (C3)/Control-senofilcon A (C3) | Control-senofilcon A (C3)/ Test-senofilcon A (C3)
Started | 91 | 90
Completed | 91 | 88
Not Completed | 0 | 2
Not completed — Unsatisfactory Lens Fitting due to Study Lens | 0 | 1
Not completed — Other: Incorrect Study Lens Dispensed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 176
  Multiple | 1
  Asian | 3
  Black or African American | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 188

OUTCOME MEASURES:

1. Primary Outcome: Distance Monocular logMAR Visual Acuity
Description: Distance Monocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast condition. Visual acuity is assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test-senofilcon A (C3): Subjects that wore the Test lens during either period 1 or period 2 of the study
- Control-senofilcon A (C3): Subjects that wore the Control lens during either period 1 or period 2 of the study
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 180 | 181
Number analyzed (Eyes) | 360 | 362
logMAR | -0.107 (0.0740) | -0.104 (0.0705)
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); It was calculated using a 1-sided one sample mean t-test with a type I error rate of 0.025 that 9 subjects provide at least 99% statistical power to test for superiority; Test type: Superiority — A superiority margin of 0.0 logMAR was used; Linear Mixed Model; Least-Square Mean = -0.13, 95% CI 1-sided [upper limit -0.10], Standard Error of Mean 0.012

2. Primary Outcome: CLUE Vision Score
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 180 | 181
Units on a scale | 68.75 (21.547) | 70.18 (19.912)
Statistical Analysis 1: Comparison: Test-senofilcon A (C3) vs Control-senofilcon A (C3); It was calculated using a 1-sided one sample mean t-test with a type I error rate of 0.025 that 165 subjects provide at least 99% statistical power to test for superiority; Test type: Superiority — A superiority margin of 62 points was used; Linear Mixed Model; Least-quares mean = 69.4, 95% CI 1-sided [lower limit 65.2], Standard Error of Mean 2.13

3. Primary Outcome: Proportion of Eyes With Absolute Rotation Less Than or Equal to 10 Degrees
Description: Absolute rotation was assessed for each subject eye using a slit lamp 15-minutes after lens insertion. Acceptable absolute rotation was dichotomized into a binary response where Y=1 if absolute rotation was less than or equal to 10 degrees and Y=0 otherwise (absolute rotation greater than 10 degrees). The proportion of eyes with absolute rotation less than or equal to 10 degrees was report for each lens.
Time Frame: 15-minutes after lens insertion
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 185 | 184
Number analyzed (Eyes) | 370 | 368
Proportion of eyes | 0.9784 | 0.9918
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.99 and an intraclass correlation of 0.70, that 100 subjects were required to test for superiority to achieve a minimum statistical power of 99% with 95% central posterior credible interval; Test type: Superiority — A superiority margin of 0.80 was used; Bayesian beta- binomial model; Method used is Bayesian beta- binomial model for correlated binary data; Mean Central Posterior Proportion = 0.974, 95% CI 2-sided [0.950 to 0.989], Standard Deviation 0.0100

4. Primary Outcome: Proportion of Eyes With Rotational Stability Less Than or Equal to 5 Degrees
Description: Rotational Stability was assessed for each subject eye using a slit lamp 15-minutes after lens insertion. Rotational Stability was dichotomized into a binary response where Y=1 if Rotational Stability was less than or equal to 5 degrees and Y=0 otherwise (Rotational Stability greater than 5 degrees). The proportion of eyes with Rotational Stability less than or equal to 5 degrees was report for each lens.
Time Frame: 15-minutes after lens insertion
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 185 | 184
Number analyzed (Eyes) | 370 | 368
Proportion of eyes | 1 | 1
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); [analysis description as in outcome 3, analysis 1]; Test type: Superiority — A superiority margin of 0.80 was used; Bayesian beta-binomial model; Method used is Bayesian beta- binomial model for correlated binary data; Mean Central Posterior Proportion = 0.989, 95% CI 2-sided [0.976 to 0.997], Standard Deviation 0.0054

5. Primary Outcome: Proportion of Eyes With Acceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion at the 1-week follow-up. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with acceptable lens fit was reported for each lens.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 185 | 184
Number analyzed (Eyes) | 370 | 368
Proportion of eyes | 1 | 1
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); [analysis description as in outcome 3, analysis 1]; Test type: Superiority — A superiority margin of 0.80 was used; Bayesian beta- binomial model; Method used is Bayesian beta- binomial model for correlated binary data; Mean Central Posterior Proportion = 0.989, 95% CI 2-sided [0.977 to 0.997], Standard Deviation 0.0053

6. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported for each lens.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 185 | 184
Number analyzed (Eyes) | 370 | 368
Proportion of eyes | 0 | 0
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.01 and an intraclass correlation of 0.70, that 100 subjects were required to test for superiority to achieve a minimum statistical power of 99% with 95% central posterior credible Interval; Test type: Superiority — A superiority margin of 0.05 was used; Bayesian beta-binomial model; Bayesian beta- binomial model for correlated binary data; Mean Central Posterior Proportion = 0.003, 95% CI 2-sided [0.000 to 0.010], Standard Deviation 0.0028

7. Secondary Outcome: CLUE Comfort Score
Description: Subjective comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score was reported.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 180 | 181
Units on a scale | 66.20 (24.134) | 67.04 (22.269)
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); It was calculated using a 1-sided one sample mean t-test with a type I error rate of 0.025 that 135 subjects provide at least 97% statistical power to test for superiority; Test type: Superiority — A superiority margin of 58 points was used; Linear Mixed Model; Least-squares Mean = 66.1, 95% CI 1-sided [lower limit 61.2], Standard Error of Mean 2.48

8. Secondary Outcome: CLUE Handling Score
Description: Subjective handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE handling score was reported.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
Number analyzed (Participants) | 180 | 181
Units on a scale | 70.30 (20.999) | 70.87 (22.752)
Statistical Analysis 1: Comparison: Test-senofilcon A (C3); [analysis description as in outcome 7, analysis 1]; Test type: Superiority — A superiority margin of 61 points was used; Linear Mixed Model; Least-squares Mean = 69.9, 95% CI 1-sided [lower limit 66.6], Standard Error of Mean 1.66

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 21 days.
Description: All subjects dispensed a study lens.
Groups:
- Test-senofilcon A (C3): Subjects that wore the Test lens during any point of the study.
- Control-senofilcon A (C3): Subjects that wore the Control lens during any point of the study.
Arm/Group | Test-senofilcon A (C3) | Control-senofilcon A (C3)
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/184
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/184
Other Adverse Events (participants affected / at risk) | 0/185 | 0/184

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT05778786/Prot_SAP_002.pdf